CLINICAL TRIAL: NCT00375856
Title: An Investigation of Computer-Assisted Total Knee Replacement Kinematics on Patient Performance: An Examination of the DePuy P.F.C.® SigmaTM Posterior Cruciate Substituting Knee and the DePuy P.F.C.® Sigma RP Rotating Platform Knee Systems
Brief Title: Computer-Assisted Total Knee Replacement Kinematics: DePuy Sigma Posterior Cruciate Substituting Knee and the DePuy Sigma RP Rotating Platform Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Dr. John Rudan, Principal Investigator, Queen's University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: DepuyRP06
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2013-05

CONDITIONS: Osteoarthritis, Knee
Keywords: arthroplasty; knee; computer-assist; gait; Total knee arthroplasty; knee prostheses
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): DePuy P.F.C.® SigmaTM Posterior Cruciate Substituting Knee
- 2 (Experimental): Rotating Platform Knee
  Interventions: Device: DePuy P.F.C.® Sigma Rotating Platform Knee

INTERVENTIONS:
Device: DePuy P.F.C.® Sigma Rotating Platform Knee — no details
  Other Names: no other name
  Arms: 2

SUMMARY:
Primary Research Questions:

1. Do patients with knee osteoarthritis (OA) who undergo total knee replacement with a Sigma rotating platform have better clinical outcomes at 2 years post surgery (i.e. quality of life, function, range of motion) than similar patients who undergo total knee arthroplasty (TKA) using the Sigma fixed bearing knee?
2. Do patients with knee OA who undergo TKA with a Sigma rotating platform have different knee kinetics and kinematics as measured by gait analysis than similar patients who undergo TKA using the Sigma fixed bearing knee?
3. Do patients with knee OA who undergo TKA with or without computer assistance have better clinical outcomes at two years following surgery (quality of life, function, range of motion)?
4. Do patients with knee OA who undergo TKA with or without computer assistance have different knee kinematics and kinetics as measured by gait analysis?

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 years
* Undergoing primary total knee arthroplasty
* Clinically significant osteoarthritic degeneration

Exclusion Criteria:

* Active articular infections
* Bilateral knee replacement (simultaneous)
* Previous joint infections
* Significant concurrent ipsilateral hip osteoarthritis
* Chronic pain syndrome requiring medications for control
* History of chemical addiction
* Significant spinal stenosis, significant symptomatic sciatica
* Patients who are unlikely to comply with, participate in, or return for follow-up visits as described in the protocol
* Osteomyelitis, septicemia or other infections that may spread to other areas of the body
* Highly communicable diseases, immuno-compromising conditions and/or conditions that may limit follow-up (eg. AIDS, active tuberculosis, venereal disease, active hepatitis, neoplastic disease)
* Decreased mental comprehension and literacy
* Prior high tibial osteotomy
* Prior patellectomy
* Rheumatoid arthritis
* Pregnancy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2006-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Gait and radiographic parameters | 0

SECONDARY OUTCOMES:
Knee pain, function | 0

CONTACTS AND LOCATIONS:
Overall Officials: John F Rudan, MD, Principal Investigator — Queen's University/Kingston General Hospital; Steve MacDonald, MD, Principal Investigator — London Health Sciences Center; Eric Bohm, MD, Principal Investigator — University of Manitoba/Concordia Hospital
Locations (3):
- Canada (3):
  - University of Manitoba, Winnipeg, Manitoba
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Center, London, Ontario